CLINICAL TRIAL: NCT00003376
Title: Phase III Trial of Methotrexate, Vinblastine, Doxorubicin and Cisplatin vs Carboplatin and Paclitaxel in Advanced Carcinoma of the Urothelium
Brief Title: Two-Drug Combination Chemotherapy Compared With Four-Drug Combination Chemotherapy in Treating Patients With Advanced Cancer of the Urothelium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066368; E4897; CLB-99908; GUMC-01011
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Cisplatin; Doxorubicin; Methotrexate; Paclitaxel; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: paclitaxel
Drug: vinblastine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if four-drug combination chemotherapy is more effective than two-drug combination chemotherapy in treating advanced cancer of the urothelium.

PURPOSE: Randomized phase III trial to compare the effectiveness of four-drug combination chemotherapy with that of two-drug combination chemotherapy in treating patients who have advanced cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the objective response rate, duration of remission, overall survival, and quality of life of patients with progressing regional or metastatic transitional cell carcinoma (or mixed histologies with a component of transitional cell carcinoma) of the urothelium treated with methotrexate, vinblastine, doxorubicin, and cisplatin vs carboplatin and paclitaxel. II. Compare the relative toxic effects of these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive methotrexate IV on days 1, 15, and 22; vinblastine IV on days 2, 15, and 22; and cisplatin IV over 2 hours and doxorubicin IV on day 2. Treatment repeats every 28 days for a total of 6 courses in the absence of unacceptable toxicity or disease progression. Arm II: Patients receive paclitaxel IV over 3 hours immediately followed by carboplatin IV over 30 minutes. Treatment repeats every 21 days for a total of 6 courses in the absence of unacceptable toxicity or disease progression. Quality of life is assessed before treatment, before courses 2 and 4, at 4 weeks after last course, and at 10 months. Patients are followed every 3 months for 1 year and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 330 patients will be accrued for this study within 3.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed transitional cell carcinoma of the urothelium (renal pelvis, ureter, bladder, or urethra) or mixed histologies containing a component of transitional cell carcinoma of the urothelium with manifestations of progressing regional or metastatic cancer Clinically unsuspected organ-confined prostate cancer found during cystoprostatectomy allowed Evaluable or measurable disease No significant pericardial or pleural effusion or edema No significant ascites No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST no greater than 2 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No history of severe cardiovascular disease (American Heart Association class III or IV), uncontrolled congestive heart failure, or cardiac dysrhythmias Other: Prior malignancy allowed if curatively treated with no evidence of recurrence No active infection requiring parenteral antibiotics Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior systemic biologic response modifier therapy No concurrent filgrastim (G-CSF) within 24 hours prior to and after study chemotherapy administration Chemotherapy: No prior systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior pelvic radiotherapy as a component of bladder-sparing therapy or as an adjuvant for locally advanced disease with positive margins No concurrent local radiotherapy for pain control or life-threatening situations Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 1998-12-03 (Actual); Primary Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Roth, MD, Study Chair — Vanderbilt-Ingram Cancer Center; Martin J. Edelman, MD, Study Chair — Veterans Affairs Medical Center - Baltimore
Locations (50):
- United States (50):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Dreicer R, Manola J, Roth BJ, See WA, Kuross S, Edelman MJ, Hudes GR, Wilding G. Phase III trial of methotrexate, vinblastine, doxorubicin, and cisplatin versus carboplatin and paclitaxel in patients with advanced carcinoma of the urothelium. Cancer. 2004 Apr 15;100(8):1639-45. doi: 10.1002/cncr.20123. PMID 15073851
- [Result] Dreicer R, Manola J, Roth B, et al.: ECOG 4897: phase III trial of methotrexate, vinblastine, doxorubicin, and cisplatin (M-VAC) versus carboplatin and paclitaxel in patients with advanced carcinoma of the urothelium. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1542, 2003.